CLINICAL TRIAL: NCT04114539
Title: A Multicenter, Open-Label, Extension Study Intended to Evaluate the Long-term Safety of Ecopipam Tablets in Children and Adolescent Subjects With Tourette's Syndrome
Brief Title: Ecopipam Tablets to Study Tourette Syndrome in Children and Adolescents - Open Label Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBS-101-OL-001
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-11

CONDITIONS: Tourette Syndrome in Children; Tourette Syndrome in Adolescence
Keywords: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — ecopipam

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ecopipam (Experimental)
  Interventions: Drug: Ecopipam

INTERVENTIONS:
Drug: Ecopipam — Ecopipam HCl 12.5-, 37.5-. 50-, 75- and 100-mg tablets; 2 mg/kg/day target dose; oral administration daily in evenings.

SUMMARY:
This study was an international, multicenter, open-label, long term extension study evaluating the safety of ecopipam tablets for the treatment of children and adolescent subjects with Tourette Syndrome.

DETAILED DESCRIPTION:
This was an international, multicenter, open-label, long term extension study to evaluate the safety of ecopipam tablets for the treatment of pediatric subjects (aged ≥6 to ≤18 years at Baseline) with Tourette Syndrome. Participants who completed the Phase 2b, randomized, double-blind, efficacy and safety study (EBS-101-CL-001) without major reportable protocol deviations, and who met all the inclusion/exclusion criteria for this study were eligible to participate in this study. All participants were titrated to a target dose of 2 mg/kg/day as participants rolled over from the Phase 2b double-blind efficacy and safety study were tapered off study drug to maintain the blind from that study. Participants were to complete study visits every month for 1 year. Follow-up visits were conducted 7 and 14 days after the last dose of the study drug and a follow-up phone call was conducted 30 days after the last dose of study drug

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed the EBS-101-CL-001 study through the Day 14 Follow Up Visit within the last 30 days (or longer with permission of the medical monitor) without a major reportable protocol deviation and must be someone the Investigator feels would benefit from continued participation.

Exclusion Criteria:

* Certain mood or psychiatric disorders (i.e., dementia, bipolar disorder, schizophrenia, major depressive disorder).
* Unstable medical illness or clinically significant lab abnormalities.
* Risk of suicide.
* Pregnant or lactating women.
* Moderate to severe renal insufficiency.
* Positive urine drug screen.
* Certain medications that would lead to drug interactions.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (53):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Advanced Research Center Inc., Anaheim, California
  - UCLA, Los Angeles, California
  - PCSD-Feighner Research, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Yale School of Medicine, New Haven, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - Northwest Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Research in Miami Inc., Hialeah, Florida
  - University of Miami, Miami, Florida
  - MedBio Trials, North Miami, Florida
  - APG Research LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Pediatric Neurology, PA, Winter Park, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Hospitals, Chicago, Illinois
  - AMR - Baber Research Inc., Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Helen DeVos Children's Hospital / Spectrum Health Medical Group, Wyoming, Michigan
  - St. Charles Psychiatric Associates dba Midwest Research Group, Saint Charles, Missouri
  - Movement Disorders Center, St Louis, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Clinical Research Center of NJ, Voorhees Township, New Jersey
  - New York Neurology Associates P.C, New York, New York
  - Hapworth Research Inc., New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Mood Disorders Consulting Medicine PLLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Quest Therapeutics of Avon Lake, Avon Lake, Ohio
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - North Star Medical Research LLC, Middleburg Heights, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Clinical Trials LLC, Bellaire, Texas
  - Relaro Medical Trials, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Road Runner Research Ltd., San Antonio, Texas
  - Noetic Psychiatry, Springville, Utah
  - University of Virginia, Charlottesville, Virginia
  - Eastside Therapeutic Resource Inc dba Core Clinical Research, Everett, Washington
- Canada (3):
  - The Kids Clinic Inc, Ajax, Ontario
  - Center for Pediatric Excellence, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- CHU Poitiers, Poitiers, France
- Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida, Germany
- Poland (7):
  - Gdanskie Centrum Zdrowia Sp z o.o., Gdansk
  - Centrum Bada Klinicznych PI-House Sp. z o.o., Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Wojewdzki Specjalistyczny Szpital Dziecicy im. sw. Ludwika w Krakowie, Krakow
  - Med-Polonia Sp. z o. o., Poznan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 sites in United States, Canada and Poland from 4 October 2019 (first participant first visit) to 11 November 2022 (last participant last visit).
Pre-assignment Details: A total of 124 participants who completed the open-labelled study EBS-101-CL-001 (NCT04007991) and who met the inclusion/exclusion criteria for this study were enrolled in the current study and received study treatment. Of the 124 enrolled participants, 121 participants were included in the modified ITT (mITT) Set and Safety Set.
Groups:
- Ecopipam HCl 2 mg/kg/Day: Participants received ecopipam hydrochloride (HCl) tablets at a targeted dose of 2 milligram per kilogram per day (mg/kg/day), orally, once daily for up to 52 weeks.
Period: Overall Study
Arm/Group | Ecopipam HCl 2 mg/kg/Day
Started | 124
Safety Set (Treated) (The Safety Set included all participants who received at least one dose of study drug from the open labelled study.) | 121
Modified Intention-to-Treat Set (The Modified Intention-to-Treat (mITT) set included all participants who received at least one dose of study drug and had at least one post Baseline scoring of Yale Global Tic Severity Scale (YGTSS).) | 121
Completed | 80
Not Completed | 44
Not completed — Adverse Event | 14
Not completed — Lost to Follow-up | 2
Not completed — Non-compliance with Protocol | 2
Not completed — Non-compliance with Study Drug | 1
Not completed — Withdrawal by Parent/Caregiver | 8
Not completed — Withdrew consent | 10
Not completed — Others not specified | 5
Not completed — Investigator Decision | 2

BASELINE CHARACTERISTICS:
Population: The mITT set included all participants who received at least one dose of study drug and had at least one post baseline scoring of YGTSS.
Groups:
- Ecopipam HCI 2 mg/kg/Day: Participants received ecopipam HCl tablets at a targeted dose of 2 mg/kg/day, orally, once daily for up to 52 weeks.
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 107
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 110
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6
  United States | 91
  Poland | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) and Their Relationship (Unrelated, Possibly Related, or Probably Related)
Description: An AE was any untoward medical condition that occurs in a participant while participating in this clinical study. It can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study. An SAE was any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. The relationship of the study drug in causing or contributing to the AE whether unrelated, possibly related, or probably related was decided by investigator medical judgment.
Time Frame: From start of study drug administration until 30 days after last dose (Up to Month 13)
Population: The Safety Set included all participants who received at least one dose of study drug from the open labelled study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 121
Participants
  Participants with any AEs | 84
  Participants with SAEs | 2
  Participants with unrelated AEs | 44
  Participants with possibly related AEs | 27
  Participants with probably related AEs | 13
  Participants with unrelated SAEs | 1
  Participants with possibly related SAEs | 1
  Participants with probably related SAEs | 0

2. Primary Outcome: Change From Baseline in Hematology Parameters: Basophils to Leukocytes Ratio Reported in Percentage of Cells
Description: Basophils/Leukocytes was measured in percentages (%). Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in basophils to leukocytes ratio is reported in terms of percentage of cells.
Time Frame: Baseline up to Month 12
Population: The Safety Set included all participants who received at least one dose of study drug from the open labelled study. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
percentage of cells | -0.1 (0.91)

3. Primary Outcome: Change From Baseline in Hematology Parameters: Eosinophils to Leukocytes Ratio Reported in Percentage of Cells
Description: Eosinophils/Leukocytes was measured in percentages (%). Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in eosinophils to leukocytes ratio is reported in terms of percentage of cells.
Time Frame: Baseline up to Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
percentage of cells | 0.1 (1.52)

4. Primary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in hematology parameter erythrocytes was reported.
Time Frame: Baseline up to Month 12
Population: The Safety Set included all participants who received at least one dose of study drug from the open labelled study. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
10^12 cells per liter | 0.04 (0.263)

5. Primary Outcome: Change From Baseline in Hematology Parameters: Hematocrit
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in hematology parameter hematocrit was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liter of cells per liter of blood (L/L)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
liter of cells per liter of blood (L/L) | 0.01 (0.029)

6. Primary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in hematology parameter hemoglobin was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmoL/L)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 38
millimoles per liter (mmoL/L) | 0.08 (0.429)

7. Primary Outcome: Change From Baseline in Hematology Parameters: Leukocytes and Platelets
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in hematology parameters (Leukocytes and Platelets) expressed in 10^9 cells per liter were reported.
Time Frame: Baseline up to Month 12
Population: The Safety Set included all participants who received at least one dose of study drug from the open labelled study. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
10^9 cells per liter
  Leukocytes | 0.15 (1.349)
  Platelets | 4.1 (51.49)

8. Primary Outcome: Change From Baseline in Hematology Parameters: Lymphocytes to Leukocytes Ratio Reported in Percentage of Cells
Description: Lymphocytes/leukocytes was measured in percentages (%). Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in lymphocytes to leukocytes ratio is reported in terms of percentage of cells.
Time Frame: Baseline up to Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
percentage of cells | 0.2 (10.20)

9. Primary Outcome: Change From Baseline in Hematology Parameters: Monocytes to Leukocytes Ratio Reported in Percentage of Cells
Description: Monocytes/leukocytes was measured in percentages (%). Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in monocytes to leukocytes ratio is reported in terms of percentage of cells.
Time Frame: Baseline up to Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
percentage of cells | 0.2 (1.43)

10. Primary Outcome: Change From Baseline in Hematology Parameters: Neutrophils to Leukocytes Ratio Reported in Percentage of Cells
Description: Neutrophils/leukocytes was measured in percentages (%). Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in neutrophils to leukocytes ratio is reported in terms of percentage of cells.
Time Frame: Baseline up to Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 37
percentage of cells | -0.3 (10.45)

11. Primary Outcome: Change From Baseline in Serum Chemistry Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Lactase Dehydrogenase
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in Serum chemistry parameters (alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, and lactate dehydrogenase) were reported.
Time Frame: Baseline up to Month 12
Population: The Safety Set included all participants who received at least one dose of study drug from the open labelled study. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "Number Analyzed" signifies participants who were evaluable at the specified categories.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 29
units per liter (U/L)
  Alanine Aminotransferase | 2.3 (9.41)
  Alkaline Phosphatase | -4.7 (80.71)
  Aspartate Aminotransferase | -0.3 (5.48)
  Lactase Dehydrogenase: number analyzed (Participants) | 26
  Lactase Dehydrogenase | -6.2 (33.96)

12. Primary Outcome: Change From Baseline in Serum Chemistry Parameters: Albumin, Globulin and Protein
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in Serum chemistry parameters (albumin, globulin and protein) were reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 29
grams per liter (g/L)
  Albumin | 0.6 (2.87)
  Globulin | 1.2 (2.92)
  Protein | 1.9 (4.63)

13. Primary Outcome: Change From Baseline in Serum Chemistry Parameters: Bicarbonate, Calcium, Chloride, Cholesterol, Glucose, Phosphate, Potassium, Sodium, Triglyceride and Urea Nitrogen
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in Serum chemistry parameters (bicarbonate, calcium, chloride, cholesterol, glucose, phosphate, potassium, sodium, triglyceride, urea nitrogen) expressed in millimoles per liter (mmol/L) were reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 29
millimoles per liter (mmol/L)
  Bicarbonate | -0.6 (3.57)
  Calcium | 0.02 (0.153)
  Chloride | -0.2 (2.54)
  Cholesterol | 0.20 (0.704)
  Glucose | -0.06 (0.781)
  Phosphate | -0.02 (0.294)
  Potassium | 0.02 (0.684)
  Sodium | -0.1 (2.22)
  Triglyceride | -0.09 (0.625)
  Urea Nitrogen | -0.07 (1.176)

14. Primary Outcome: Change From Baseline in Serum Chemistry Parameters: Bilirubin, Creatinine and Direct Bilirubin
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in Serum chemistry parameters (bilirubin, creatinine and direct bilirubin) expressed in micromole per liter (mcmol/L) were reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 29
mcmol/L
  Bilirubin: number analyzed (Participants) | 26
  Bilirubin | -0.6 (4.78)
  Creatinine | 6.2 (8.85)
  Direct Bilirubin: number analyzed (Participants) | 28
  Direct Bilirubin | -0.1 (0.77)

15. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured to identify average blood glucose concentration over prolonged periods of time. Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in HbA1c was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 30
percentage of HbA1c | 0.03 (0.313)

16. Primary Outcome: Change From Baseline in Vital Signs Parameter: Diastolic Blood Pressure and Systolic Blood Pressure
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in vital signs parameters diastolic blood pressure and systolic blood pressure and according to the assessment position (supine and standing) expressed in millimeter(s) of mercury (mmHg) was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 75
mmHg
  Diastolic Blood Pressure: number analyzed (Participants) | 74
  Diastolic Blood Pressure | 0.9 (9.96)
  Diastolic Blood Pressure: Supine: number analyzed (Participants) | 74
  Diastolic Blood Pressure: Supine | 0.6 (8.58)
  Diastolic Blood Pressure: Standing | 1.6 (10.65)
  Systolic Blood Pressure: number analyzed (Participants) | 74
  Systolic Blood Pressure | 0.3 (11.47)
  Systolic Blood Pressure: Supine: number analyzed (Participants) | 74
  Systolic Blood Pressure: Supine | 1.8 (11.35)
  Systolic Blood Pressure: Standing | -1.1 (12.15)

17. Primary Outcome: Change From Baseline in Vital Signs Parameter: Pulse Rate
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in vital sign parameter pulse rate and according to assessment position (supine and standing) was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 75
beats per minute (bpm)
  Pulse Rate: number analyzed (Participants) | 74
  Pulse Rate | 0.4 (13.76)
  Pulse Rate Supine: number analyzed (Participants) | 74
  Pulse Rate Supine | 0.6 (14.20)
  Pulse Rate Standing | 1.8 (18.09)

18. Primary Outcome: Change From Baseline in Vital Signs Parameter: Body Mass Index [BMI]
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in vital signs parameter BMI was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 75
kilograms per square meter (kg/m^2) | 1.0 (4.58)

19. Primary Outcome: Change From Baseline in Vital Signs Parameter: Height
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in vital signs height was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 75
centimeter (cm) | 4.0 (3.90)

20. Primary Outcome: Change From Baseline in Vital Signs Parameter: Weight
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change from baseline in vital signs parameter weight was reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 75
kilogram (kg) | 5.4 (13.53)

21. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Values Parameters: Aggregate PR Interval, Aggregate QRS Duration, Aggregate QT Interval, and Aggregate QTc Interval
Description: Baseline was defined as the last measurement taken before the first dose of open-label treatment on Day 1 of current study. Change From Baseline in ECG parameters aggregate PR interval, aggregate QRS duration, aggregate QT interval, and aggregate QTc interval expressed in millisecond (msec) was reported.
Time Frame: Baseline to Month 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 73
millisecond (msec)
  Aggregate PR interval | -5.6 (18.81)
  Aggregate QRS duration | -0.6 (9.76)
  Aggregate QT interval | 5.5 (30.26)
  Aggregate QTc interval | 0.2 (38.53)

22. Primary Outcome: Number of Participants With Clinically Significant Abnormal Physical Examination Findings
Description: Physical examination included examination of the following body areas and systems: Head, Eyes, Ears, Nose, Mouth, Throat, Neck (including Thyroid), Thorax, Abdomen, Urogenital, Extremities, Neurological, Skin and Mucosae and Others. Any clinically significant abnormalities in physical examination were judged by the investigator. Only non-zero values are reported.
Time Frame: Baseline up to Month 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 74
Participants
  Neurological | 1
  Other: number analyzed (Participants) | 1
  Other | 1

23. Secondary Outcome: Change From Baseline in the Yale Global Tic Severity Scale -Total Tic Score (YGTSS-TTS) at Months 1, 3, 6, 9 and 12
Description: The YGTSS was a clinician-completed rating scale used to quantify overall tic severity as well as specific subdomains of tic number, frequency, intensity, complexity and interference. Each of these subdomains was scored, on a 0 to 5 scale, separately for motor and vocal tics and then summed across both motor and vocal tics to yield a total tic score ranging from 0 to 50. Higher scores represent more severe symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline up to Months 1, 3, 6, 9 and 12
Population: The mITT set included all participants who received at least one dose of study drug and had at least one post Baseline scoring of YGTSS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "Number Analyzed" signifies participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 119
score on a scale
  Change at Month 1 | -6.5 (7.10)
  Change at Month 3: number analyzed (Participants) | 114
  Change at Month 3 | -7.5 (8.04)
  Change at Month 6: number analyzed (Participants) | 99
  Change at Month 6 | -10.6 (8.88)
  Change at Month 9: number analyzed (Participants) | 91
  Change at Month 9 | -11.5 (8.34)
  Change at Month 12: number analyzed (Participants) | 81
  Change at Month 12 | -11.7 (9.48)

24. Secondary Outcome: Change From Baseline in the Yale Global Tic Severity Scale - Impairment (YGTSS-I) at Months 1, 3, 6, 9 and 12
Description: The YGTSS was a clinician-completed rating scale used to quantify overall tic severity as well as specific subdomains of tic number, frequency, duration, intensity, and complexity. Each of these subdomains was scored, on 0 to 5 scale, separately for an overall impairment rating from (0 = ''none'' to 50 = ''severe''). Higher score represent more severe symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline up to Months 1, 3, 6, 9 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 119
score on a scale
  Change at Month 1 | -7.2 (9.74)
  Change at Month 3: number analyzed (Participants) | 114
  Change at Month 3 | -8.3 (10.88)
  Change at Month 6: number analyzed (Participants) | 99
  Change at Month 6 | -10.4 (10.49)
  Change at Month 9: number analyzed (Participants) | 91
  Change at Month 9 | -12.5 (11.11)
  Change at Month 12: number analyzed (Participants) | 81
  Change at Month 12 | -12.1 (11.59)

25. Secondary Outcome: Change From Baseline in the Yale Global Tic Severity Scale - Global Score (YGTSS-GS) at Months 1, 3, 6, 9 and 12
Description: The YGTSS was a clinician-completed rating scale used to quantify overall tic severity as well as specific subdomains of tic number, frequency, duration, intensity, and complexity. Each of these subdomains was scored, on a 0 to 5 scale, separately for motor and vocal tics and then summed across both motor and vocal tics to yield a tic severity score ranging from 0 to 50. The YGTSS also provides for an overall impairment rating (0 = ''none'' to 50 = ''severe''). YGTSS-GS is the total of YGTSS-TTS and YGTSS-I. The maximum YGTSS Global score is 100, while the maximum motor score is 25, the maximum vocal score is 25, and the maximum impairment score is 50. Higher scores indicate more severe tics. A negative change from baseline indicates improvement.
Time Frame: Baseline up to Months 1, 3, 6, 9 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 119
score on a scale
  Change at Month 1 | -13.8 (15.07)
  Change at Month 3: number analyzed (Participants) | 114
  Change at Month 3 | -15.9 (16.91)
  Change at Month 6: number analyzed (Participants) | 99
  Change at Month 6 | -21.0 (17.64)
  Change at Month 9: number analyzed (Participants) | 91
  Change at Month 9 | -24.0 (17.31)
  Change at Month 12: number analyzed (Participants) | 81
  Change at Month 12 | -23.8 (19.11)

26. Secondary Outcome: Change From Baseline in Clinical Global Impression of Tourette Syndrome of Severity (CGI-TS-S) at Months 1, 3, 6, 9, 12
Description: The CGI consists of 2 reliable and valid 7-item Likert scales used to assess severity and change in clinical symptoms. The CGI severity scale (CGI-TS-S) ranges from 1 = "not ill at all" to 7 = "among the most extremely ill." Higher scores represent more severe symptoms. A negative change from baseline indicates improvement.
Time Frame: Baseline up to Months 1, 3, 6, 9, 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 119
score on a scale
  Change at Month 1 | -0.8 (1.02)
  Change at Month 3: number analyzed (Participants) | 114
  Change at Month 3 | -0.8 (1.10)
  Change at Month 6: number analyzed (Participants) | 99
  Change at Month 6 | -1.0 (1.10)
  Change at Month 9: number analyzed (Participants) | 91
  Change at Month 9 | -1.2 (1.13)
  Change at Month 12: number analyzed (Participants) | 81
  Change at Month 12 | -1.2 (1.21)

27. Secondary Outcome: Clinical Global Impression Tourette Syndrome of Improvement (CGI-TS-I) Scores at Months 1, 3, 6, 9 and 12
Description: The CGI consists of 2 reliable and valid 7-item Likert scales used to assess severity and change in clinical symptoms. The scale ranges from 1 = "very much improved" to 7 = very much worse" for the CGI-TS-I. Higher score represent more severe symptoms.
Time Frame: Months 1, 3, 6, 9 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 120
score on a scale
  Month 1 | 2.7 (1.05)
  Month 3: number analyzed (Participants) | 114
  Month 3 | 2.5 (1.24)
  Month 6: number analyzed (Participants) | 99
  Month 6 | 2.2 (1.04)
  Month 9: number analyzed (Participants) | 91
  Month 9 | 2.0 (1.02)
  Month 12: number analyzed (Participants) | 81
  Month 12 | 2.0 (1.09)

28. Secondary Outcome: Change From Baseline in Gilles de la Tourette Syndrome-Quality of Life Scale for Children and Adolescents (C&A-GTS-QOL) Total Score at Months 1, 3, 6, 9 and 12
Description: The C&A-GTS-QOL was a 27-item questionnaire specific to TS patients that asks the patient to assess the extent to which their quality of life is impacted by their symptoms. The C&A-GTS-QOL consists of 6 subscales (cognitive [score range 0-32], coprophenomena [range 0-12], psychological [range 0-24], physical [range 0-12], obsessive-compulsive [range 0-16], and activities of daily living (ADL) [range 0-12] and uses a 5 point Likert scale ranging from no problem to extreme problem. Scores for six subscales were generated by summing items and, for ease of interpretation, transformation to a range of 0 to 100 (100* [(observed score-min possible score)/(max possible score-min possible score)]). Total score, resulted from sum of the subscale scores, was also normalized to a 0 to 100 range. Higher score indicated worst quality of life. A negative change from baseline indicates better quality of life.
Time Frame: Baseline up to Months 1, 3, 6, 9 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ecopipam HCI 2 mg/kg/Day
Number analyzed (Participants) | 117
score on a scale
  Change at Month 1 | -4.0 (11.30)
  Change at Month 3: number analyzed (Participants) | 114
  Change at Month 3 | -4.5 (12.30)
  Change at Month 6: number analyzed (Participants) | 98
  Change at Month 6 | -7.7 (13.97)
  Change at Month 9: number analyzed (Participants) | 91
  Change at Month 9 | -6.7 (16.91)
  Change at Month 12: number analyzed (Participants) | 80
  Change at Month 12 | -8.0 (16.17)

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after last dose of the study drug (Up to Month 13)
Arm/Group | Ecopipam HCI 2 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 2/121
Other Adverse Events (participants affected / at risk) | 84/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ecopipam HCI 2 mg/kg/Day (N=121)
Abdominal pain upper (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Obsessive thoughts (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecopipam HCI 2 mg/kg/Day (N=121)
Tourette's disorder (Congenital, familial and genetic disorders) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vision blurred (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (10)
Nausea (Gastrointestinal disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Tooth impacted (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2)
Tooth resorption (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 7 (9)
Fatigue (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 17 (28)
Upper respiratory tract infection (Infections and infestations) | 7 (7)
COVID-19 (Infections and infestations) | 6 (6)
Influenza (Infections and infestations) | 4 (4)
Rhinitis (Infections and infestations) | 4 (8)
Pharyngitis (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
Adenoiditis (Infections and infestations) | 1 (1)
Body tinea (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (3)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 1 (1)
Testicular injury (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Hepatic enzyme increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (9)
Somnolence (Nervous system disorders) | 8 (8)
Dizziness (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (4)
Migraine (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Akathisia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Formication (Nervous system disorders) | 1 (1)
Narcolepsy (Nervous system disorders) | 1 (1)
Postural tremor (Nervous system disorders) | 1 (1)
Tongue biting (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 11 (12)
Insomnia (Psychiatric disorders) | 9 (9)
Depression (Psychiatric disorders) | 5 (8)
Tic (Psychiatric disorders) | 5 (6)
Aggression (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Depressed mood (Psychiatric disorders) | 2 (2)
Depressive symptom (Psychiatric disorders) | 2 (2)
Dissociative disorder (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1)
Bruxism (Psychiatric disorders) | 1 (1)
Compulsions (Psychiatric disorders) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Social anxiety disorder (Psychiatric disorders) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 1 (1)
Terminal insomnia (Psychiatric disorders) | 1 (2)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Vein collapse (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must consult their clinical trial agreement. In summary, PI shall have the right to publish, present or otherwise use the results for their research publication objectives, provided that such Publication does not disclose Confidential Information. PI shall submit in writing to Sponsor any material at least 90 days for review and comment. Sponsor shall advise PI of any information which is Confidential Information or which may impair Sponsor's ability to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT04114539/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04114539/SAP_001.pdf